CLINICAL TRIAL: NCT04482179
Title: A Phase II, Randomized, Blinded Study of Transcranial Magnetic Stimulation and Constraint Induced Language Therapy for the Treatment of Chronic Aphasia - Alzheimer Disease Sub-study
Brief Title: Transcranial Magnetic Stimulation and Constraint Induced Language Therapy for Alzheimer Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, H. Branch Coslett, Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 831532; R01DC016800-01A1 (NIH)
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either TMS or sham TMS in a 2:1 allocation ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The individual administering TMS will keep the master file of subject assignments, but all other individuals in contact with the subject or their data will be unaware of group assignment. Participants will not be informed of their assignment to active or sham status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TMS (Active Comparator): There will be 10 TMS sessions over 2 consecutive weeks in which 30 two-second stimulation trains of 10 Hz TMS will be delivered every 30 seconds to the left inferior pars triangularis and to the left posterior superior left temporal gyrus. Each TMS treatment session will be immediately followed by a 60-90 minute session of Constrained Induced Language Therapy (CILT).
  Interventions: Device: Active TMS; Behavioral: CILT
- Sham TMS (Sham Comparator): There will be 10 TMS sessions over 2 consecutive weeks in which 30 two-second stimulation trains of 10 Hz sham TMS will be delivered every 30 seconds to the left inferior pars triangularis and to the left posterior superior left temporal gyrus. Sham TMS will be administered with a sham TMS coil that looks and sounds like the active coil but does not generate a magnetic field. Each TMS treatment session will be immediately followed by a 60-90 minute session of Constrained Induced Language Therapy (CILT).
  Interventions: Behavioral: CILT; Device: Sham TMS

INTERVENTIONS:
Device: Active TMS — Active TMS will be delivered at 100% motor threshold
  Arms: Active TMS
Behavioral: CILT — 60-90 minutes of CILT will be administered during each treatment session
  Other Names: Constraint Induced Language Therapy
Device: Sham TMS — Sham TMS will be administered
  Arms: Sham TMS

SUMMARY:
Impaired verbal communication is a cardinal symptom of Alzheimer Disease (AD) and the source of enormous distress and disability. Effective therapies for this deficit are lacking. In light of the emerging literature demonstrating that Transcranial Magnetic Stimulation (TMS) improves general cognition in subjects with Alzheimer Disease (AD), the investigators propose to study the effectiveness of TMS as a therapy for impaired verbal communication. The hypothesis to be tested is that TMS combined with Constraint Induced Language Therapy (CILT) improves verbal communication more than sham TMS and CILT. A second aim is to use state-of-the-art neuroimaging to understand the mechanisms underlying any beneficial effect of the treatment.

DETAILED DESCRIPTION:
TMS is a technique by which a brief electrical current is induced in brain tissue causing a brief suppression of the excitability of the underlying tissue; the technique, which was introduced in the 1980s and has been extensively used around the world, has been shown to transiently improve or disrupt specific cognitive operations. To achieve this end, a coil is positioned against the subject's head. The delivery of a single pulse begins with the discharge of current from a capacitor into a circular or figure-of-eight coil; this electrical current generates a brief magnetic field of up to 2.2 Tesla. As the pulse of electricity has a rise time of 0.2 ms. and a duration of 1 ms., the magnetic field changes in intensity quite rapidly. Because the magnetic field passes freely through the scalp, skull, and meninges, the flux in the magnetic field induces a small electric field in the brain that transiently alters neural activity.

TMS may be delivered in a variety of ways. The investigators propose to use 10 Hz TMS; that is, TMS pulses will be delivered at a frequency of 10/second, for a total of 1200 pulses. Using the figure-of-eight coil to be employed here, TMS is thought to affect activity in approximately 1 cubic cm. of cortex. Many investigators have employed TMS for AD with a frequency of 10 Hz and most have delivered 1200 pulses per session.

The baseline phase will consist of 3 sessions, each lasting 1-2 hours depending on the stamina of the subject. The point of the baseline testing is to characterize the subject's language function. To that end, a number of standard language and neuropsychological tasks will be administered. These include the Western Aphasia Battery, Pyramids and Palm Trees test, Figural Fluency Test, word and non-word repetition tasks, spontaneous narrative production, CILT stimulus naming, and the Repeatable Battery for the Assessment of Neuropsychological Status. Additionally, during the baseline, subjects will undergo MRI of the brain or, if they have a contraindication to MRI, a CAT scan of the head. No contrast will be used.

In the treatment phase, there will be 10 TMS sessions over 2 consecutive weeks in which 30 two-second stimulation trains of 10 Hz TMS will be delivered every 30 seconds to the left inferior pars triangularis and to the left posterior superior left temporal gyrus at 100% motor threshold. There will be a total of 600 pulses to each site in each session for a total of 1200 pulses per session. Each TMS treatment session will be immediately followed by a 60-90 minute session of CILT.

There will be two 3-month post-treatment visits and two 6-month post-treatment visits in which the full battery of language and cognitive assessments will be repeated. Subjects who are able to undergo MRI scanning will have anatomic and fMRI scans at the first 6-month post-treatment visit.

The investigators will pair TMS with CILT which has been shown to have positive outcomes in post-stroke aphasia. CILT invokes use-dependent learning in communicative interactions by requiring spoken output and restricting use of alternative forms of communication, such as gestures. The investigators will use a dual card-matching task modeled after Maher et al. As in the original CILT design, the participant interacts verbally with a conversational partner (here, the speech language pathologist), in turn requesting a card of given description and complying with the partner's request. In this way, the treatment targets both production and comprehension. Moreover, as verbal targets increase in linguistic complexity across the protocol ("a ball", "throw a ball"; "Do you have a ball"?), a variety of lexical and phrasal structures are targeted. Studies of CILT have reported gains on multiple language behaviors, supporting its broad engagement of the language network.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of mild-moderate AD as defined by the National Institute of Aging - Alzheimer's Disease and Related Disorders Association criteria
* Mild-moderate cognitive impairment, indicated by Mini-Mental Status Exam (MMSE) scores between 23 and 15 inclusive
* Must be right handed as defined by the Edinburgh Handedness Inventory
* Must be a native English speaker
* Must be able to understand the nature of the study, and give informed consent

Exclusion Criteria:

* History of stroke
* History of seizure
* History of any other significant neurologic disease (e.g., ALS)
* Significant depression as defined by the Geriatric Depression Scale.
* Any significant medical disorder that, in the view of the investigators, could threaten the subject's ability to complete the study (e.g., cancer, significant cardiac disease)
* Any contraindications to TMS, including uncontrolled seizures, previous brain surgery, and history of tinnitus

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Branch Coslett, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamilton RH, Chrysikou EG, Coslett B. Mechanisms of aphasia recovery after stroke and the role of noninvasive brain stimulation. Brain Lang. 2011 Jul;118(1-2):40-50. doi: 10.1016/j.bandl.2011.02.005. Epub 2011 Apr 2. PMID 21459427
- [Background] Medina J, Norise C, Faseyitan O, Coslett HB, Turkeltaub PE, Hamilton RH. Finding the Right Words: Transcranial Magnetic Stimulation Improves Discourse Productivity in Non-fluent Aphasia After Stroke. Aphasiology. 2012 Sep 1;26(9):1153-1168. doi: 10.1080/02687038.2012.710316. Epub 2012 Aug 29. PMID 23280015
- [Background] Seniow J, Waldowski K, Lesniak M, Iwanski S, Czepiel W, Czlonkowska A. Transcranial magnetic stimulation combined with speech and language training in early aphasia rehabilitation: a randomized double-blind controlled pilot study. Top Stroke Rehabil. 2013 May-Jun;20(3):250-61. doi: 10.1310/tsr2003-250. PMID 23841973
- [Background] Silvanto J, Muggleton N, Walsh V. State-dependency in brain stimulation studies of perception and cognition. Trends Cogn Sci. 2008 Dec;12(12):447-54. doi: 10.1016/j.tics.2008.09.004. Epub 2008 Oct 24. PMID 18951833
- [Background] Ayache SS, Farhat WH, Zouari HG, Hosseini H, Mylius V, Lefaucheur JP. Stroke rehabilitation using noninvasive cortical stimulation: motor deficit. Expert Rev Neurother. 2012 Aug;12(8):949-72. doi: 10.1586/ern.12.83. PMID 23002939
- [Background] Kakuda W, Abo M, Shimizu M, Sasanuma J, Okamoto T, Yokoi A, Taguchi K, Mitani S, Harashima H, Urushidani N, Urashima M; NEURO Investigators. A multi-center study on low-frequency rTMS combined with intensive occupational therapy for upper limb hemiparesis in post-stroke patients. J Neuroeng Rehabil. 2012 Jan 20;9(1):4. doi: 10.1186/1743-0003-9-4. PMID 22264239
- [Background] Koganemaru S, Mima T, Thabit MN, Ikkaku T, Shimada K, Kanematsu M, Takahashi K, Fawi G, Takahashi R, Fukuyama H, Domen K. Recovery of upper-limb function due to enhanced use-dependent plasticity in chronic stroke patients. Brain. 2010 Nov;133(11):3373-84. doi: 10.1093/brain/awq193. Epub 2010 Aug 5. PMID 20688810
- [Background] Shewan CM, Kertesz A. Reliability and validity characteristics of the Western Aphasia Battery (WAB). J Speech Hear Disord. 1980 Aug;45(3):308-24. doi: 10.1044/jshd.4503.308. PMID 7412225
- [Background] Mirman D, Chen Q, Zhang Y, Wang Z, Faseyitan OK, Coslett HB, Schwartz MF. Neural organization of spoken language revealed by lesion-symptom mapping. Nat Commun. 2015 Apr 16;6:6762. doi: 10.1038/ncomms7762. PMID 25879574
- [Background] Howard, D., & Patterson, K. E. (1992). The Pyramids and Palm Trees Test: A Test of Semantic Access from Words and Pictures. Thames Valley Test Company
- [Background] Nicholas LE, Brookshire RH. A system for quantifying the informativeness and efficiency of the connected speech of adults with aphasia. J Speech Hear Res. 1993 Apr;36(2):338-50. doi: 10.1044/jshr.3602.338. PMID 8487525
- [Background] Foygel, D., & Dell, G. S. (2000). Models of impaired lexical access in speech production. Journal of Memory and Language, 43(2), 182-216.
- [Background] Pulvermuller F, Neininger B, Elbert T, Mohr B, Rockstroh B, Koebbel P, Taub E. Constraint-induced therapy of chronic aphasia after stroke. Stroke. 2001 Jul;32(7):1621-6. doi: 10.1161/01.str.32.7.1621. PMID 11441210
- [Background] Medaglia JD, Huang W, Segarra S, Olm C, Gee J, Grossman M, Ribeiro A, McMillan CT, Bassett DS. Brain network efficiency is influenced by the pathologic source of corticobasal syndrome. Neurology. 2017 Sep 26;89(13):1373-1381. doi: 10.1212/WNL.0000000000004324. Epub 2017 Aug 4. PMID 28779011
- [Background] Ahmed MA, Darwish ES, Khedr EM, El Serogy YM, Ali AM. Effects of low versus high frequencies of repetitive transcranial magnetic stimulation on cognitive function and cortical excitability in Alzheimer's dementia. J Neurol. 2012 Jan;259(1):83-92. doi: 10.1007/s00415-011-6128-4. Epub 2011 Jun 14. PMID 21671144
- [Background] Bentwich J, Dobronevsky E, Aichenbaum S, Shorer R, Peretz R, Khaigrekht M, Marton RG, Rabey JM. Beneficial effect of repetitive transcranial magnetic stimulation combined with cognitive training for the treatment of Alzheimer's disease: a proof of concept study. J Neural Transm (Vienna). 2011 Mar;118(3):463-71. doi: 10.1007/s00702-010-0578-1. Epub 2011 Jan 19. PMID 21246222
- [Background] Brem, A. K., Schilberg, L., Freitas, C., Atkinson, N., Seligson, E., & Pascual-Leone, A. (2013). Effects of cognitive training and rTMS in Alzheimer's disease. Alzheimer's & Dementia: The Journal of the Alzheimer's Association, 9(4), P664.
- [Background] Buckner RL, Sepulcre J, Talukdar T, Krienen FM, Liu H, Hedden T, Andrews-Hanna JR, Sperling RA, Johnson KA. Cortical hubs revealed by intrinsic functional connectivity: mapping, assessment of stability, and relation to Alzheimer's disease. J Neurosci. 2009 Feb 11;29(6):1860-73. doi: 10.1523/JNEUROSCI.5062-08.2009. PMID 19211893
- [Background] Cheng CPW, Wong CSM, Lee KK, Chan APK, Yeung JWF, Chan WC. Effects of repetitive transcranial magnetic stimulation on improvement of cognition in elderly patients with cognitive impairment: a systematic review and meta-analysis. Int J Geriatr Psychiatry. 2018 Jan;33(1):e1-e13. doi: 10.1002/gps.4726. Epub 2017 May 11. PMID 28493371
- [Background] Cotelli M, Calabria M, Manenti R, Rosini S, Zanetti O, Cappa SF, Miniussi C. Improved language performance in Alzheimer disease following brain stimulation. J Neurol Neurosurg Psychiatry. 2011 Jul;82(7):794-7. doi: 10.1136/jnnp.2009.197848. Epub 2010 Jun 23. PMID 20574108
- [Background] Cotelli M, Manenti R, Cappa SF, Geroldi C, Zanetti O, Rossini PM, Miniussi C. Effect of transcranial magnetic stimulation on action naming in patients with Alzheimer disease. Arch Neurol. 2006 Nov;63(11):1602-4. doi: 10.1001/archneur.63.11.1602. PMID 17101829
- [Background] Deters KD, Nho K, Risacher SL, Kim S, Ramanan VK, Crane PK, Apostolova LG, Saykin AJ; Alzheimer's Disease Neuroimaging Initiative. Genome-wide association study of language performance in Alzheimer's disease. Brain Lang. 2017 Sep;172:22-29. doi: 10.1016/j.bandl.2017.04.008. Epub 2017 May 31. PMID 28577822
- [Background] Drumond Marra HL, Myczkowski ML, Maia Memoria C, Arnaut D, Leite Ribeiro P, Sardinha Mansur CG, Lancelote Alberto R, Boura Bellini B, Alves Fernandes da Silva A, Tortella G, Ciampi de Andrade D, Teixeira MJ, Forlenza OV, Marcolin MA. Transcranial Magnetic Stimulation to Address Mild Cognitive Impairment in the Elderly: A Randomized Controlled Study. Behav Neurol. 2015;2015:287843. doi: 10.1155/2015/287843. Epub 2015 Jun 16. PMID 26160997
- [Background] Engels MM, Stam CJ, van der Flier WM, Scheltens P, de Waal H, van Straaten EC. Declining functional connectivity and changing hub locations in Alzheimer's disease: an EEG study. BMC Neurol. 2015 Aug 20;15:145. doi: 10.1186/s12883-015-0400-7. PMID 26289045
- [Background] Faroqi-Shah, Y., & Virion, C. R. (2009). Constraint-induced language therapy for agrammatism: Role of grammaticality constraints. Aphasiology, 23(7-8), 977-988.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Fornito A, Zalesky A, Breakspear M. The connectomics of brain disorders. Nat Rev Neurosci. 2015 Mar;16(3):159-72. doi: 10.1038/nrn3901. PMID 25697159
- [Background] Haffen E, Chopard G, Pretalli JB, Magnin E, Nicolier M, Monnin J, Galmiche J, Rumbach L, Pazart L, Sechter D, Vandel P. A case report of daily left prefrontal repetitive transcranial magnetic stimulation (rTMS) as an adjunctive treatment for Alzheimer disease. Brain Stimul. 2012 Jul;5(3):264-266. doi: 10.1016/j.brs.2011.03.003. Epub 2011 Mar 30. No abstract available. PMID 22037125
- [Background] Hameister, I., Nickels, L., Abel, S., & Croot, K. (2017). "Do you have mowing the lawn?"-improvements in word retrieval and grammar following constraint-induced language therapy in primary progressive aphasia. Aphasiology, 31(3), 308-331.
- [Background] Hodges JR, Salmon DP, Butters N. Semantic memory impairment in Alzheimer's disease: failure of access or degraded knowledge? Neuropsychologia. 1992 Apr;30(4):301-14. doi: 10.1016/0028-3932(92)90104-t. PMID 1603295
- [Background] Koch G, Bonni S, Pellicciari MC, Casula EP, Mancini M, Esposito R, Ponzo V, Picazio S, Di Lorenzo F, Serra L, Motta C, Maiella M, Marra C, Cercignani M, Martorana A, Caltagirone C, Bozzali M. Transcranial magnetic stimulation of the precuneus enhances memory and neural activity in prodromal Alzheimer's disease. Neuroimage. 2018 Apr 1;169:302-311. doi: 10.1016/j.neuroimage.2017.12.048. Epub 2017 Dec 19. PMID 29277405
- [Background] Lee J, Choi BH, Oh E, Sohn EH, Lee AY. Treatment of Alzheimer's Disease with Repetitive Transcranial Magnetic Stimulation Combined with Cognitive Training: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study. J Clin Neurol. 2016 Jan;12(1):57-64. doi: 10.3988/jcn.2016.12.1.57. Epub 2015 Sep 11. PMID 26365021
- [Background] Martin A, Fedio P. Word production and comprehension in Alzheimer's disease: the breakdown of semantic knowledge. Brain Lang. 1983 May;19(1):124-41. doi: 10.1016/0093-934x(83)90059-7. PMID 6860932
- [Background] Medaglia JD, Lynall ME, Bassett DS. Cognitive network neuroscience. J Cogn Neurosci. 2015 Aug;27(8):1471-91. doi: 10.1162/jocn_a_00810. Epub 2015 Mar 24. PMID 25803596
- [Background] Mohs RC, Rosen WG, Davis KL. The Alzheimer's disease assessment scale: an instrument for assessing treatment efficacy. Psychopharmacol Bull. 1983;19(3):448-50. No abstract available. PMID 6635122
- [Background] Norise C, Hamilton RH. Non-invasive Brain Stimulation in the Treatment of Post-stroke and Neurodegenerative Aphasia: Parallels, Differences, and Lessons Learned. Front Hum Neurosci. 2017 Jan 23;10:675. doi: 10.3389/fnhum.2016.00675. eCollection 2016. PMID 28167904
- [Background] Rabey JM, Dobronevsky E. Repetitive transcranial magnetic stimulation (rTMS) combined with cognitive training is a safe and effective modality for the treatment of Alzheimer's disease: clinical experience. J Neural Transm (Vienna). 2016 Dec;123(12):1449-1455. doi: 10.1007/s00702-016-1606-6. Epub 2016 Sep 8. PMID 27631152
- [Background] Rabey JM, Dobronevsky E, Aichenbaum S, Gonen O, Marton RG, Khaigrekht M. Repetitive transcranial magnetic stimulation combined with cognitive training is a safe and effective modality for the treatment of Alzheimer's disease: a randomized, double-blind study. J Neural Transm (Vienna). 2013 May;120(5):813-9. doi: 10.1007/s00702-012-0902-z. Epub 2012 Oct 18. PMID 23076723
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rubinov M, Sporns O. Complex network measures of brain connectivity: uses and interpretations. Neuroimage. 2010 Sep;52(3):1059-69. doi: 10.1016/j.neuroimage.2009.10.003. Epub 2009 Oct 9. PMID 19819337
- [Background] Saur D, Lange R, Baumgaertner A, Schraknepper V, Willmes K, Rijntjes M, Weiller C. Dynamics of language reorganization after stroke. Brain. 2006 Jun;129(Pt 6):1371-84. doi: 10.1093/brain/awl090. Epub 2006 Apr 25. PMID 16638796
- [Background] Stam CJ. Modern network science of neurological disorders. Nat Rev Neurosci. 2014 Oct;15(10):683-95. doi: 10.1038/nrn3801. Epub 2014 Sep 4. PMID 25186238
- [Background] Szatloczki G, Hoffmann I, Vincze V, Kalman J, Pakaski M. Speaking in Alzheimer's Disease, is That an Early Sign? Importance of Changes in Language Abilities in Alzheimer's Disease. Front Aging Neurosci. 2015 Oct 20;7:195. doi: 10.3389/fnagi.2015.00195. eCollection 2015. PMID 26539107
- [Background] Vacas SM, Stella F, Loureiro JC, Simoes do Couto F, Oliveira-Maia AJ, Forlenza OV. Noninvasive brain stimulation for behavioural and psychological symptoms of dementia: A systematic review and meta-analysis. Int J Geriatr Psychiatry. 2019 Sep;34(9):1336-1345. doi: 10.1002/gps.5003. Epub 2018 Oct 17. PMID 30246461
- [Background] van den Heuvel MP, Hulshoff Pol HE. Exploring the brain network: a review on resting-state fMRI functional connectivity. Eur Neuropsychopharmacol. 2010 Aug;20(8):519-34. doi: 10.1016/j.euroneuro.2010.03.008. Epub 2010 May 14. PMID 20471808
- [Background] van den Heuvel MP, Sporns O. Network hubs in the human brain. Trends Cogn Sci. 2013 Dec;17(12):683-96. doi: 10.1016/j.tics.2013.09.012. PMID 24231140
- [Background] Wu Y, Xu W, Liu X, Xu Q, Tang L, Wu S. Adjunctive treatment with high frequency repetitive transcranial magnetic stimulation for the behavioral and psychological symptoms of patients with Alzheimer's disease: a randomized, double-blind, sham-controlled study. Shanghai Arch Psychiatry. 2015 Oct;27(5):280-8. doi: 10.11919/j.issn.1002-0829.215107. PMID 26977125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2019-2021 from the Hospital of the University of Pennsylvania and surrounding Philadelphia area medical centers.
Pre-assignment Details: A total of 11 participants did not qualify at the time of enrollment due to MMSE scores (8) and medical contraindication (3).
  One participant dropped out of the study prior to randomization due to travel concerns.
Groups:
- Active TMS: Participants will receive 10 TMS sessions over 2 consecutive weeks in which 20 minutes of TMS will be delivered to the left inferior pars triangularis and to the left posterior superior left temporal gyrus.
  Each TMS treatment session will be immediately followed by a 60-90 minute session of Constrained Induced Language Therapy (CILT).
- Sham TMS: Participants will take part in 10 sham TMS sessions over 2 consecutive weeks. Sham TMS mimics the sensory experience (look, sound and feel) of active TMS but does not stimulate the brain. Sham TMS will be administered with a sham TMS coil that looks and sounds like the active coil but does not generate a magnetic field. The sham TMS will target the same two brain locations - left inferior pars triangularis and the left posterior superior left temporal gyrus.
  Each sham TMS treatment session will be immediately followed by a 60-90 minute session of Constrained Induced Language Therapy (CILT).
Period: Overall Study
Arm/Group | Active TMS | Sham TMS
Started | 7 | 4
Completed | 5 | 4
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS | Sham TMS | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (3.66) | 73.4 (1.76) | 71.27 (3.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 2 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Western Aphasia Battery (WAB-AQ) Score [Mean (Standard Deviation); unit: scores on a scale] | 80.7 (7.8) | 87.4 (6.1) | 83.1 (7.7)
Philadelphia Naming Test, Items Correct [Mean (Standard Deviation); unit: number of items correct] | 121.0 (37.6) | 157.3 (15.5) | 134.2 (35.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in WAB-AQ Score
Description: The primary outcome measure will be the change in score on the Western Aphasia Battery Aphasia Quotient (WAB-AQ), a score assessing overall aphasia recovery. Scores can range from 0-100, with higher scores representing better outcomes. 0-25 is very severe, 26-50 is severe, 51-75 is moderate, and 76-above is mild. A score of 93 or higher is considered recovered.
Time Frame: 12 weeks post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 5 | 4
score on a scale | -1.7 (4.3) | -.1 (7.3)
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; Test type: Superiority; p < .05, Regression, Linear

2. Secondary Outcome: Change in Percentage of Items Correct on the PNT
Description: The secondary outcome measure will be change in naming accuracy on the Philadelphia Naming Test (PNT). PNT naming accuracy is measured as a percentage from 0% to 100% with higher percentages meaning better naming ability. The task involves naming 175 pictures of common objects.
Time Frame: 12 weeks post-treatment
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 5 | 4
percentage of correct responses | -3.2 (8.2) | -5.0 (6.1)
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; Test type: Superiority; p < .05, Regression, Linear

ADVERSE EVENTS:
Time Frame: From baseline, adverse event data were collected over a period of time consisting of 12 weeks.
Description: Adverse event (AEs) information was collected daily during treatment sessions, as well as each follow-up visit.
Arm/Group | Active TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/4
Other Adverse Events (participants affected / at risk) | 2/7 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=7) | Sham TMS (N=4)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) — Participant died from cardiac arrest.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=7) | Sham TMS (N=4)
Headache (General disorders) | 2 (4) | 1 (3)
Head Pain (General disorders) | 1 (1) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (2)
Stomach Ache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heart Palpitations (Cardiac disorders) | 0 (0) | 1 (2)
Fall (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT04482179/Prot_SAP_000.pdf